CLINICAL TRIAL: NCT05538793
Title: Deep Learning for the Discrimination Among Bacterial, Fungal, Viral, Amebic and Noninfectious Keratitis: a Nationwide Study
Brief Title: Deep Learning for the Discrimination Among Different Types of Keratits: a Nationwide Study
Status: Completed | Type: Observational
Sponsor: Ningbo Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEH2022091015
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Keratitis; Automatic Judgement; Image
Keywords: Keratitis; Slit-lamp Image; Deep Learning
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detecting the cause of keratitis fast is the premise of providing targeted therapy for reducing vision loss and preventing severe complications. Due to overlapping inflammatory features, even expert cornea specialists have relatively poor performance in the identification of causative pathogen of infectious keraitis. In this project, the investigators aim to develop an automated and accurate deep learning system to discriminate among bacterial, fungal, viral, amebic and noninfectious keratitis based on slit-lamp images and evaluated this system using the datasets obtained from mutiple independent clinical centers across China.

ELIGIBILITY:
Inclusion Criteria:

Slit-lamp images with sufficient diagnostic certainty and showing keratitis at the active phase.

Exclusion Criteria:

* Poor-quality images
* Images presenting mixed infections (i.e., cornea infected by two or more causative pathogens)

Ages: 1 Week to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Child, Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 10369 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve of the deep learning system | 2020-2022

SECONDARY OUTCOMES:
Accuracy of the deep learning system | 2020-2022
Sensitivity of the deep learning system | 2020-2022
Specificity of the deep learning system | 2020-2022

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ningbo Eye Hospital, Ningbo, Zhejiang
  - Eye Hospital of Wenzhou Medical University, Wenzhou